CLINICAL TRIAL: NCT06900075
Title: Efficacy and Safety of Efsubaglutide Alfa Injection 3 Mg Every Two Weeks in Patients with Type 2 Diabetes: a Multicenter, Randomized, Open-Label Study
Brief Title: Efficacy and Safety of Efsubaglutide Alfa Injection 3 Mg Q2W in T2D Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Yinnuo Pharmaceutical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YN011-304
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Efsubaglutide Alfa 3 mg Q2W-1 mg QW (Experimental)
  Interventions: Drug: Efsubaglutide Alfa 3mg Q2W and 1mg QW
- Efsubaglutide Alfa 1 mg QW-3 mg Q2W (Active Comparator)
  Interventions: Drug: Efsubaglutide Alfa 1mg QW and 3mg Q2W

INTERVENTIONS:
Drug: Efsubaglutide Alfa 3mg Q2W and 1mg QW — Efsubaglutide Alfa 3 mg administered once every two weeks for 8 weeks, followed by a switch to Efsubaglutide Alfa 1 mg administered once weekly for an additional 8 weeks of treatment.
  Arms: Efsubaglutide Alfa 3 mg Q2W-1 mg QW
Drug: Efsubaglutide Alfa 1mg QW and 3mg Q2W — Efsubaglutide Alfa 1 mg administered once weekly for 8 weeks, followed by a switch to Efsubaglutide Alfa 3 mg administered once every two weeks for an additional 8 weeks of treatment.
  Arms: Efsubaglutide Alfa 1 mg QW-3 mg Q2W

SUMMARY:
This study is a multicenter, randomized, open-label, active-controlled clinical trial with a two-period crossover design, aimed at evaluating the efficacy and safety of Efsubaglutide Alfa Injection 3 mg administered Q2W in patients with Type 2 Diabetes Mellitus (T2DM) who have inadequate glycemic control despite dietary and exercise interventions. The primary endpoint is time in range (TIR; glucose concentration 3·9-10·0 mmol/L) during the period from Week 6 to Week 8 of Efsubaglutide Alfa Injection treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years (inclusive) at screening, with no restriction on gender;
2. Diagnosed with Type 2 Diabetes Mellitus (T2DM) according to the 2024 ADA 3.Diabetes Management Standards for at least 8 weeks prior to screening, and no antidiabetic treatment received within the 8 weeks prior to screening;

4.Glycated Hemoglobin (HbA1c) between ≥7.5% and ≤11.0% at screening; 5.Fasting Plasma Glucose (FPG) ≤13.9 mmol/L at screening; 6.Body Mass Index (BMI) between 19.0 and 35.0 kg/m² (inclusive) at screening; 7.Subjects must be able to understand the purpose and content of the study, willing to receive relevant treatments, voluntarily participate in the study, and provide written informed consent.

Exclusion Criteria:

1. Patients with Type 1 diabetes or other specific types of diabetes;
2. Receipt of any of the following medications or treatments: a. Use of antidiabetic medications (including herbal medicines, other traditional medicines, and health products) within 2 months prior to screening; b. Use of non-antidiabetic medications that may significantly affect glucose metabolism for ≥7 days within 2 months prior to screening [e.g., glucocorticoids (excluding inhaled, ophthalmic, or topical applications), growth hormones, sympathomimetic agents (e.g., isoproterenol, dopamine, atropine), high-dose salicylates (e.g., aspirin >300 mg/day), danazol, octreotide, or anabolic androgenic steroids (e.g., oxymetholone, oxandrolone)].
3. Presence of any of the following medical histories or conditions: a. Known hypersensitivity to glucagon-like peptide-1 (GLP-1) receptor agonists; b. History of diabetic ketoacidosis, hyperglycemic hyperosmolar state, or lactic acidosis within 6 months prior to screening; c. Presence of unstable or treatment-requiring proliferative retinopathy or maculopathy, severe diabetic neuropathy, intermittent claudication, or diabetic foot within 6 months prior to screening; d. Severe hypoglycemia (Grade 3) events within 6 months prior to screening, or non-severe hypoglycemia occurring 3 or more times within 1 month prior to screening; e. History of gastroparesis, or clinically significant gastric emptying abnormalities, or severe gastrointestinal diseases as deemed by the investigator; f. Presence of any condition that may cause hemolysis or erythrocyte instability affecting HbA1c measurements (e.g., hematologic malignancies, hemolytic anemia, sickle cell disease); g. History of acute or chronic pancreatitis; h. History of acute cholecystitis within 6 months prior to screening, or symptomatic or treatment-requiring cholelithiasis within 6 months prior to screening (except for subjects who have undergone cholecystectomy and are clinically stable); i. Presence of Cushing's syndrome, hyperthyroidism, or inadequately controlled hypothyroidism at screening (except for subjects who have subclinical hypothyroidism not requiring thyroid hormone therapy as determined by the investigator and with TSH <10 mIU/ml); j. History of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma, or a family history of these conditions in a first-degree relative; k. Presence of the following cardiovascular or cerebrovascular conditions within 6 months prior to screening: decompensated heart failure (NYHA Class III or IV), treatment-requiring arrhythmia, unstable angina or myocardial infarction, coronary artery bypass grafting or percutaneous coronary intervention, stroke (ischemic or hemorrhagic), or transient ischemic attack; l. History of malignancy within the past 5 years (excluding clinically cured cervical carcinoma in situ or basal cell carcinoma of the skin) or potential malignancy under evaluation; m. Severe trauma, severe infection, or surgery that may affect glycemic control within 1 month prior to screening, or planned surgery that may interfere with study completion or compliance.
4. Presence of any of the following conditions at screening or prior to randomization: a. Sitting systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg; b. Clinically relevant abnormalities on a 12-lead electrocardiogram (ECG) that may affect subject safety or interpretation of study results (e.g., treatment-requiring arrhythmia); c. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5×ULN, or total bilirubin (TBIL) >2.0×ULN; d. Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m² (using CKD-EPI formula); e. Serum calcitonin ≥50 ng/L (pg/mL); f. Hemoglobin <100 g/L; g. Fasting triglycerides ≥5.7 mmol/L; h. Serum amylase and/or lipase ≥3×ULN.
5. Presence of the following serological abnormalities at screening: a. Positive HIV antibody; b. Positive hepatitis C antibody (HCV-Ab); c. Positive syphilis-specific antibody; d. Positive hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb); if either test is positive, HBV-DNA quantification must be performed, and subjects with results ≥ the lower limit of detection are excluded from the study.
6. Receipt of blood or plasma products within 3 months prior to screening, or blood donation or blood loss exceeding 400 mL within 3 months prior to screening.
7. Known or suspected history of alcohol abuse within the past year [defined as a weekly alcohol intake greater than 14 units (1 unit = approximately 360 mL of beer, 45 mL of spirits with 40% alcohol, or 150 mL of wine)].
8. History of drug abuse or substance dependence.
9. Pregnant or breastfeeding women at screening, or those with a positive pregnancy test.
10. Subjects of childbearing potential (or female partners of male subjects) who intend to conceive from the time of informed consent signing until 3 months after the last dose, or who are unwilling to use effective contraceptive measures.
11. Participation in other clinical trials with investigational drugs within 3 months prior to screening.
12. Any other conditions deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Time in range (TIR) | 6-8 weeks
  The primary endpoint is time in range (TIR; glucose concentration 3·9-10·0 mmol/L) during the period from Week 6 to Week 8 of Efsubaglutide Alfa Injection treatment.

SECONDARY OUTCOMES:
Glycated Albumin (GA) | 8 weeks
TIR | 6-8 weeks
  Change in TIR From Baseline
Time in tight range (TTIR) | 6-8 weeks
  TTIR is defined as the percentage of time that glucose readings are within 3·9-7·8 mmol/L
Time above range (TAR) | 6-8 weeks
Time below range (TBR) | 6-8 weeks
Glucose Management Indicator (GMI) | 6-8 weeks
Coefficient of variation (CV) | 6-8 weeks
Standard deviation of blood glucose (SDBG) | 6-8 weeks
Mean amplitude of glycemic excursions (MAGE) | 6-8 weeks
HbA1c | 8 weeks